CLINICAL TRIAL: NCT01854697
Title: A Randomized, Open-Label Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 and ABT-333 Co-administered With and Without Ribavirin Compared to Telaprevir Co-administered With Pegylated Interferon α-2a and Ribavirin in Treatment-Naïve Adults With Chronic Hepatitis C Genotype 1 Virus Infection (MALACHITE I)
Brief Title: A Study to Evaluate the Efficacy and Safety of Three Experimental Drugs Compared With Telaprevir (a Licensed Product) in People With Hepatitis C Virus Infection Who Have Not Had Treatment Before
Acronym: MALACHITE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-774; 2012-003754-84 (EudraCT Number)
Record Dates: First submitted 2013-04-08; First posted 2013-05-15 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-07

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic Hepatitis C; Interferon Free; Hepatitis C Treatment Naive; Hepatitis C Virus; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — dasabuvir; Viekira Pak; ombitasvir; paritaprevir; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A: 3-DAA + RBV in GT1a (Experimental): ABT-450/r/ABT-267 150 mg/100 mg/25 mg once daily (QD) and ABT-333 250 mg twice daily (BID) and weight-based RBV for 12 weeks (3 direct-acting antivirals [DAAs] with RBV in GT1a)
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin
- Arm B: TPV/PR in GT1a (Active Comparator): Telaprevir (TPV) 750 mg every 8 hours (q8h) and pegIFN 180 µg/week and weight-based RBV (PR) for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight-based RBV according to response guided therapy per the prescribing information for telaprevir (telaprevir with pegIFN/RBV in GT1a)
  Interventions: Drug: Ribavirin; Drug: Telaprevir; Drug: Pegylated Interferon alpha 2-a (PegIFN)
- Arm C: 3-DAA + RBV in GT1b (Experimental): ABT-450/r/ABT-267 150 mg/100 mg/25 mg QD and ABT-333 250 mg BID and weight-based RBV for 12 weeks (3 DAAs with RBV in GT1b)
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333; Drug: Ribavirin
- Arm D: 3-DAA in GT1b (Experimental): ABT-450/r/ABT-267 150 mg/100 mg/25 mg QD and ABT-333 250 mg BID for 12 weeks (3 DAAs without RBV in GT1b)
  Interventions: Drug: ABT-450/r/ABT-267, ABT-333
- Arm E: TPV/PR in GT1b (Active Comparator): Telaprevir 750 mg q8h and pegIFN 180 µg/week and weight-based RBV for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight-based RBV according to response guided therapy per the prescribing information for telaprevir (telaprevir with pegIFN/RBV in GT1b)
  Interventions: Drug: Ribavirin; Drug: Telaprevir; Drug: Pegylated Interferon alpha 2-a (PegIFN)

INTERVENTIONS:
Drug: ABT-450/r/ABT-267, ABT-333 — Tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: Viekira Pak; ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ABT-333 also known as dasabuvir; Holkira Pak
  Arms: Arm A: 3-DAA + RBV in GT1a; Arm C: 3-DAA + RBV in GT1b; Arm D: 3-DAA in GT1b
Drug: Ribavirin — Tablet
  Arms: Arm A: 3-DAA + RBV in GT1a; Arm B: TPV/PR in GT1a; Arm C: 3-DAA + RBV in GT1b; Arm E: TPV/PR in GT1b
Drug: Telaprevir — Film-coated tablet
  Arms: Arm B: TPV/PR in GT1a; Arm E: TPV/PR in GT1b
Drug: Pegylated Interferon alpha 2-a (PegIFN) — Pre-filled syringe
  Arms: Arm B: TPV/PR in GT1a; Arm E: TPV/PR in GT1b

SUMMARY:
This is a study to evaluate the efficacy and safety of three experimental drugs compared with telaprevir (a licensed product) in people with hepatitis C virus infection who have not had treatment before.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate that treatment with ABT-450/ritonavir (r)/ABT-267 and ABT-333 administered with or without ribavirin (RBV) has non-inferior efficacy compared to treatment with telaprevir and pegylated interferon alpha-2a (pegIFN) and RBV and to compare the safety of these regimens in treatment-naive hepatitis C virus (HCV) genotype (GT) 1a- and 1b-infected adults.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years, inclusive, at time of Screening
* Females must be post-menopausal for more than 2 years or surgically sterile or practicing abstinence/specific forms of birth control
* Subject has never received antiviral treatment for hepatitis C infection
* Chronic HCV Genotype-1 infection prior to study enrollment

Exclusion Criteria:

* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency virus antibody (HIV Ab)
* Females who are pregnant or plan to become pregnant, or breastfeeding
* Any current or past clinical evidence of cirrhosis
* Screening laboratory analyses that showing abnormal laboratory results
* Use of contraindicated medications within 2 weeks of dosing and subject with contraindication for telaprevir, pegIFN and RBV
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol
* Positive screen for drugs or alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Luo, MD, PhD, Study Director — AbbVie

REFERENCES:
- [Result] Dore GJ, Conway B, Luo Y, Janczewska E, Knysz B, Liu Y, Streinu-Cercel A, Caruntu FA, Curescu M, Skoien R, Ghesquiere W, Mazur W, Soza A, Fuster F, Greenbloom S, Motoc A, Arama V, Shaw D, Tornai I, Sasadeusz J, Dalgard O, Sullivan D, Liu X, Kapoor M, Campbell A, Podsadecki T. Efficacy and safety of ombitasvir/paritaprevir/r and dasabuvir compared to IFN-containing regimens in genotype 1 HCV patients: The MALACHITE-I/II trials. J Hepatol. 2016 Jan;64(1):19-28. doi: 10.1016/j.jhep.2015.08.015. Epub 2015 Aug 29. PMID 26321288
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: 3-DAA + RBV in GT1a: ABT-450/ritonavir (r)/ABT-267 150 mg/100 mg/25 mg once daily (QD) and ABT-333 250 mg twice daily (BID) and weight-based ribavirin (RBV) for 12 weeks (3 Direct-Acting Antivirals (DAAs) with RBV in genotype [GT] 1a)
- Arm B: TPV/PR in GT1a: Telaprevir (TPV) 750 mg every 8 hours (q8h) and pegylated interferon (pegIFN) 180 µg/week and weight-based RBV for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight based RBV according to response guided therapy per the prescribing information for telaprevir (telaprevir with pegIFN/RBV in GT1a)
- Arm E: TPV/PR in GT1b: Telaprevir 750 mg q8h and pegIFN 180 µg/week and weight-based RBV for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight based RBV according to response guided therapy per the prescribing information for telaprevir (telaprevir with pegIFN/RBV in GT1b)
Period: Overall Study
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Started | 69 | 34 | 84 | 83 | 41
Completed | 63 | 31 | 82 | 80 | 39
Not Completed | 6 | 3 | 2 | 3 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 4 | 1 | 1 | 2 | 0
Not completed — To enter another AbbVie study | 1 | 0 | 0 | 0 | 1
Not completed — Withdrew Consent | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: 3-DAA + RBV in GT1a: ABT-450/r/ABT-267 150 mg/100 mg/25 mg QD and ABT-333 250 mg BID and weight-based RBV for 12 weeks (3 DAAs with RBV in GT1a)
- Arm B: TPV/PR in GT1a: TPV 750 mg q8h and pegIFN 180 µg/week and weight-based RBV for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight based RBV according to response guided therapy per the prescribing information for telaprevir (telaprevir with pegIFN/RBV in GT1a)
- Total: Total of all reporting groups
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b | Total
Number analyzed (Participants) | 69 | 34 | 84 | 83 | 41 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (12.25) | 44.5 (14.10) | 46.2 (11.34) | 47.1 (11.33) | 45.9 (10.78) | 46.2 (11.75)
Age, Customized [Number; unit: participants]
  < 55 years | 46 | 23 | 59 | 60 | 31 | 219
  >= 55 years | 23 | 11 | 25 | 23 | 10 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 46 | 43 | 24 | 151
  Male | 48 | 17 | 38 | 40 | 17 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment (SVR12) - Primary Efficacy Analyses
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 34 | 84 | 83 | 41
percentage of participants | 97.1 | 82.4 | 98.8 | 97.6 | 78.0
Statistical Analysis 1: Comparison: Arm A: 3-DAA + RBV in GT1a vs Arm B: TPV/PR in GT1a; Test type: Non-Inferiority or Equivalence — The primary endpoint assessment comparison was made within each of the 2 HCV genotypes (GT1a and GT1b). Within HCV GT1a, the 3-DAA + RBV and TPV/PR arms were compared. Within HCV GT1b, the 3-DAA and TPV/PR arms were compared. The test treatment arm was considered noninferior to the TPV/PR arm in the respective HCV subtype if the lower bound of the 2-sided 95% CI for the treatment arm difference was above the noninferiority margin of -10.5%; Difference = 14.7, 95% CI 2-sided [1.3 to 28.2] — Difference (95% CI) from TPV/PR within GT1a. Calculated using the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Arm D: 3-DAA in GT1b vs Arm E: TPV/PR in GT1b; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 19.5, 95% CI 2-sided [6.4 to 32.6] — Difference (95% CI) from TPV/PR within GT1b. Calculated using the normal approximation to the binomial distribution

2. Secondary Outcome: Mean Change From Baseline to the Final Treatment Visit in Short-Form 36 Version 2 Health Status Survey (SF-36V2) Mental Component Summary (MCS)
Description: SF-36V2 is a generic 36-item questionnaire measuring health-related quality of life (HRQoL) covering 2 summary measures: physical component summary (PCS) and MCS; it consists of 8 subscales. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have choices per item. Scoring is done for both MCS subscale scores and summary scores; for each, the range is 0 (worst HRQoL) to 100 (best HRQoL).
Time Frame: From Day 1 of treatment up to 12 weeks for Arms A, C and D and up to 24 or 48 weeks for Arms B and E
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug and a baseline and post-baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 32 | 84 | 83 | 40
units on a scale | -4.2 (10.59) | -5.8 (12.18) | -0.3 (8.89) | -0.1 (7.73) | -6.4 (11.78)
Statistical Analysis 1: Comparison: Arm A: 3-DAA + RBV in GT1a vs Arm B: TPV/PR in GT1a; Test type: Superiority or Other; p = 0.351, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean Difference = 2.13, 95% CI 2-sided [-2.39 to 6.65], Standard Error of Mean 2.28
Statistical Analysis 2: Comparison: Arm C: 3-DAA + RBV in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean of Difference = 5.83, 95% CI 2-sided [2.19 to 9.47], Standard Error of Mean 1.84
Statistical Analysis 3: Comparison: Arm D: 3-DAA in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean of Difference = 5.28, 95% CI 2-sided [2.01 to 8.54], Standard Error of Mean 1.65

3. Secondary Outcome: Mean Change From Baseline to the Final Treatment Visit in SF-36V2 Physical Component Summary (PCS)
Description: SF-36V2 is a generic 36-item questionnaire measuring HRQoL covering 2 summary measures: PCS and MCS; it consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, bodily pain, and general health perception. Participants self-report on items in a subscale that have choices per item. Scoring is done for both PCS subscale scores and summary scores; for each, the range is 0 (worst HRQoL) to 100 (best HRQoL).
Time Frame: From Day 1 of treatment up to 12 weeks for Arms A, C and D and up to 24 or 48 weeks for Arms B and E
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 32 | 84 | 83 | 40
units on a scale | 0.5 (8.63) | -5.5 (8.26) | 0.4 (5.80) | 2.2 (4.34) | -5.5 (11.46)
Statistical Analysis 1: Comparison: Arm A: 3-DAA + RBV in GT1a vs Arm B: TPV/PR in GT1a; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean Difference = 6.08, 95% CI 2-sided [2.72 to 9.44], Standard Error of Mean 1.69
Statistical Analysis 2: Comparison: Arm C: 3-DAA + RBV in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean Difference = 6.20, 95% CI 2-sided [3.55 to 8.85], Standard Error of Mean 1.34
Statistical Analysis 3: Comparison: Arm D: 3-DAA in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included baseline score and region as covariates and treatment arm as a factor; Least Squares Mean Difference = 6.86, 95% CI 2-sided [4.36 to 9.37], Standard Error of Mean 1.27

4. Secondary Outcome: Percentage of Participants With SVR12 - Secondary Efficacy Analyses
Description: The percentage of participants with sustained virologic response (plasma HCV RNA level < LLOQ) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of active study drug
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 34 | 84 | 83 | 41
percentage of participants | 97.1 | 82.4 | 98.8 | 97.6 | 78.0
Statistical Analysis 1: Comparison: Arm A: 3-DAA + RBV in GT1a vs Arm B: TPV/PR in GT1a; Test type: Superiority or Other; p = 0.021, Regression, Logistic; Logistic regression model with treatment arm, baseline log10 HCV RNA level, and interleukin 28B (IL28B) genotype (CC versus non-CC) as predictors; Odds Ratio (OR) = 7.2, 95% CI 2-sided [1.4 to 38.0]
Statistical Analysis 2: Comparison: Arm C: 3-DAA + RBV in GT1b vs Arm E: TPV/PR in GT1b; Test type: Non-Inferiority or Equivalence — The test treatment arm was considered noninferior to the TPV/PR arm in the GT1b HCV subtype if the lower bound of the 2-sided 95% CI for the treatment arm difference was above the noninferiority margin of -10.5%; Difference = 20.8, 95% CI 2-sided [7.9 to 33.6] — Difference (95% CI) from TPV/PR within GT1b. Calculated using the normal approximation to the binomial distribution
Statistical Analysis 3: Comparison: Arm C: 3-DAA + RBV in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Calculated using logistic regression model with treatment arm, baseline log10 HCV RNA level, and IL28B genotype (CC versus non-CC) as predictors; Odds Ratio (OR) = 28.2, 95% CI 2-sided [3.3 to 241.1]
Statistical Analysis 4: Comparison: Arm D: 3-DAA in GT1b vs Arm E: TPV/PR in GT1b; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; Stratum-adjusted Cochran-Mantel-Haenszel after adjusting for IL28B genotype (CC or non-CC)

5. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: Participants in Arms A, C or D demonstrating any of the following were considered virologic failures and discontinued therapy:
  * Confirmed increase from nadir in HCV RNA (defined as 2 consecutive HCV RNA measurements of >1 log10 IU/mL above nadir) at any time point during treatment
  * Failure to achieve HCV RNA < LLOQ by Week 6 or
  * Confirmed HCV RNA ≥ LLOQ (defined as 2 consecutive HCV RNA measurements ≥ LLOQ) at any point after HCV RNA < LLOQ during treatment after HCV RNA < LLOQ.
  Participants in Arms B and E followed virologic stopping criteria described in the TPV Summary of Product Characteristics; they were considered virologic failures and discontinued therapy as follows:
  * HCV RNA > 1000 IU/mL at Week 4 to Week 12, discontinue TPV and pegIFN and RBV
  * HCV RNA > 1000 IU/mL at Week 12, discontinue pegIFN and RBV
  * Confirmed HCV RNA > lower limit of detection (LLOD) at Week 24, discontinue pegIFN and RBV
  * Confirmed HCV RNA > LLOD at Week 36, discontinue pegIFN and RBV.
Time Frame: 12 weeks for Arms A, C and D and 24 weeks or 48 weeks for Arms B and E
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 34 | 84 | 83 | 41
percentage of participants | 2.9 | 5.9 | 0 | 1.2 | 12.2

6. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Hepatitis C virus (HCV) ribonucleic acid (RNA) confirmed greater than or equal to the lower limit of quantification (LLOQ) between the end of treatment and 24 weeks post treatment among participants completing treatment and with HCV RNA less than the LLOQ at the end of treatment.
Time Frame: Within 24 weeks post treatment
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug and had sustained virologic response at Week 24 (SVR24).
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 66 | 28 | 84 | 81 | 32
percentage of participants | 0 | 0 | 1.2 | 0 | 6.3

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Treatment (SVR24)
Description: The percentage of participants with sustained virologic response (plasma HCV RNA level < LLOQ) 24 weeks after the last dose of study drug.
Time Frame: 24 weeks after the last actual dose of active study drug
Population: Intent-to-treat Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: 3-DAA + RBV in GT1a | Arm B: TPV/PR in GT1a | Arm C: 3-DAA + RBV in GT1b | Arm D: 3-DAA in GT1b | Arm E: TPV/PR in GT1b
Number analyzed (Participants) | 69 | 34 | 84 | 83 | 41
percentage of participants | 95.7 | 82.4 | 97.6 | 97.6 | 78.0
Statistical Analysis 1: Comparison: Arm A: 3-DAA + RBV in GT1a vs Arm B: TPV/PR in GT1a; Test type: Non-Inferiority or Equivalence — The test treatment arm was considered noninferior to the TPV/PR arm in the GT1a HCV subtype if the lower bound of the 2-sided 95% CI for the treatment arm difference was above the noninferiority margin of -10.5%; Difference = 13.3, 95% CI 2-sided [-0.4 to 27.0] — Difference (95% CI) from TPV/PR within GT1a. Calculated using the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Arm C: 3-DAA + RBV in GT1b vs Arm E: TPV/PR in GT1b; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 2]; Difference = 19.6, 95% CI 2-sided [6.5 to 32.7] — Difference (95% CI) from TPV/PR within GT1b. Calculated using the normal approximation to the binomial distribution
Statistical Analysis 3: Comparison: Arm D: 3-DAA in GT1b vs Arm E: TPV/PR in GT1b; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 2]; Difference = 19.5, 95% CI 2-sided [6.4 to 32.6] — Difference (95% CI) from TPV/PR within GT1b. Calculated using the normal approximation to the binomial distribution

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) collected from time of study drug administration until 30 days following discontinuation or completion of study drug administration, up to 96 weeks. Serious AEs collected from signing of informed consent until study completion.
Groups:
- 3 DAA + RBV: ABT-450/r/ABT-267 150 mg/100 mg/25 mg QD and ABT-333 250 mg BID and weight-based RBV for 12 weeks
- 3 DAA: ABT-450/r/ABT-267 150 mg/100 mg/25 mg QD and ABT-333 250 mg BID for 12 weeks
- TPV + PEGIFN + RBV: TPV 750 mg q8h and pegIFN 180 μg/week and weight-based RBV for 12 weeks followed by an additional 12 or 36 weeks of pegIFN and weight based RBV according to response guided therapy per the prescribing information for telaprevir
Arm/Group | 3 DAA + RBV | 3 DAA | TPV + PEGIFN + RBV
Serious Adverse Events (participants affected / at risk) | 1/153 | 0/83 | 9/75
Other Adverse Events (participants affected / at risk) | 100/153 | 29/83 | 74/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 DAA + RBV (N=153) | 3 DAA (N=83) | TPV + PEGIFN + RBV (N=75)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 2
RETINOPATHY (Eye disorders) | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 DAA + RBV (N=153) | 3 DAA (N=83) | TPV + PEGIFN + RBV (N=75)
ANAEMIA (Blood and lymphatic system disorders) | 10 | 1 | 32
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 14
VISION BLURRED (Eye disorders) | 0 | 1 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 1 | 6
ANAL PRURITUS (Gastrointestinal disorders) | 1 | 0 | 10
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 4
DIARRHOEA (Gastrointestinal disorders) | 15 | 7 | 12
DRY MOUTH (Gastrointestinal disorders) | 5 | 0 | 4
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 4
NAUSEA (Gastrointestinal disorders) | 32 | 7 | 30
VOMITING (Gastrointestinal disorders) | 11 | 1 | 14
ASTHENIA (General disorders) | 11 | 2 | 15
CHILLS (General disorders) | 3 | 3 | 7
FATIGUE (General disorders) | 21 | 4 | 23
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 1 | 7
INJECTION SITE ERYTHEMA (General disorders) | 0 | 0 | 5
PYREXIA (General disorders) | 4 | 2 | 16
NASOPHARYNGITIS (Infections and infestations) | 13 | 4 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 1 | 3
URINARY TRACT INFECTION (Infections and infestations) | 2 | 1 | 5
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 1 | 17
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 5
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 1 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 | 2 | 12
DIZZINESS (Nervous system disorders) | 7 | 2 | 13
DYSGEUSIA (Nervous system disorders) | 2 | 0 | 6
HEADACHE (Nervous system disorders) | 41 | 16 | 23
LETHARGY (Nervous system disorders) | 6 | 0 | 4
DEPRESSION (Psychiatric disorders) | 3 | 0 | 7
INSOMNIA (Psychiatric disorders) | 14 | 0 | 7
IRRITABILITY (Psychiatric disorders) | 11 | 0 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 1 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 1 | 10
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 19 | 5 | 26
RASH (Skin and subcutaneous tissue disorders) | 12 | 0 | 17
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.